CLINICAL TRIAL: NCT07165691
Title: TELEhealth Shared Decision-making COaching for Lung Cancer Screening in Primary Care (TELESCOPE) for Hispanics
Acronym: TELESCOPE-H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: New Jersey Commission on Cancer Research (Unknown)
Responsible Party: Principal Investigator, Evelyn Arana, DrPH, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro2025001472
Record Dates: First submitted 2025-08-26; First posted 2025-09-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lung Neoplasms
Keywords: lung cancer screening; shared decision making; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases | interventions — Telescopes

STUDY DESIGN:
Intervention Model Description: The investigators will conduct three focus groups and interviews to culturally adapt the intervention materials for a heterogeneous Hispanic population (Aim 1). After the intervention is culturally adapted, clinicians serving large numbers of Hispanic patients will be the unit of randomization (Aims 2-3). The investigators will randomize 1:1 clinicians to the culturally adapted intervention (TELESCOPE) versus enhanced usual care (EUC). Patients of clinicians will all be assigned to the arm to which the clinician was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELESCOPE intervention (Experimental): Participants will be surveyed at baseline and at one-week after the scheduled primary care office visit. If a participant is a current smoker then they are offered and navigated to evidence-based smoking cessation. If the participant is interested in screening, an LDCT is ordered. Support for screening, diagnostic testing and oncology care will be provided as needed from the Nurse Navigators.
  Interventions: Behavioral: TELESCOPE, Remote Decision Coaching with Navigation Intervention
- Enhanced Usual Care (No Intervention): Participants will be surveyed at baseline and at one-week after the scheduled primary care office visit. Primary and secondary outcome data related to the office visit will be collected.

INTERVENTIONS:
Behavioral: TELESCOPE, Remote Decision Coaching with Navigation Intervention — The TELESCOPE intervention involves three complementary components: 1) decision aid and coaching for LCS, 2) referral of current smokers to evidence-based smoking cessation services, and 3) for participants interested in screening, navigation to complete LCS and diagnostic testing and oncology care as needed
  Arms: TELESCOPE intervention

SUMMARY:
Aim 1: Culturally adapt the TELESCOPE intervention for Hispanics. Using iterative qualitative feedback from a study-specific Community Advisory Board, focus groups, and interviews with community members, the investigators will culturally adapt the TELESCOPE intervention for Hispanics at high risk for lung cancer.

Aim 2: Assess the feasibility, acceptability, and implementation potential of the culturally adapted TELESCOPE intervention delivered by bilingual patient navigators for Hispanics. Hypothesis 1: The investigators expect a recruitment rate of ≥60%, ≥90% of Hispanic participants will complete the 1-week follow-up assessments, ≥80% of the key intervention components will be delivered with 80% fidelity by the patient navigators, and ≥90% of participants and clinicians will agree or completely agree that the intervention was feasible and acceptable.

Aim 3: Explore the impact of a culturally adapted TELESCOPE intervention delivered by bilingual patient navigators vs enhanced usual care (EUC) on the initial uptake of low-dose computed tomography (LDCT) and quality of the shared decision-making (SDM) process. Hypothesis 2: The investigators expect that an adapted TELESCOPE intervention will result in higher uptake of LDCT and higher SDM quality for lung cancer screening (LCS) compared to EUC.

DETAILED DESCRIPTION:
This pilot feasibility trial aims to culturally adapt an existing TELESCOPE (R01HL158850) intervention to create a culturally appropriate SDM and navigation intervention for Hispanics in primary care settings. The investigators will assess its feasibility and acceptability (primary outcomes), and explore its impact on the uptake of LDCT (secondary outcome) compared to enhanced usual care (training clinicians to discuss LCS) for LCS in Hispanics.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 (Cultural Adaptation):

To be eligible, patients must:

1. Identify as Hispanic and/or Latino(a)
2. Able to read and speak in English or Spanish
3. Be 50 to 77 years of age
4. Be a current or former smoker
5. Have at least a 20-pack-year smoking history

Aims 2-3 (Pilot Randomized Controlled Trial)

To be eligible, patients must:

* Identify as Hispanic or Latino(a)
* Able to speak and read in English or Spanish
* Be 50 to 77 years of age
* Be a current or former smoker having quit within the past 15 years
* Have at least a 20 pack-year smoking history
* Be scheduled for a non-acute care visit at one of the study sites.
* Not coughing up blood in the last two weeks

Interviews

Providers completing the semi-structured interviews will be:

* A practicing primary care clinician or a clinic director (n=20), nursing director, or clinic practice administrator at one of the participating sites, or a TELESCOPE study patient navigator and nurse navigator
* Age 18 or older
* Fluent in English

Online surveys

Providers completing online PRISM construct surveys will be:

* A practicing primary care provider at one of the participating sites or a TELESCOPE study navigator
* Age 18 or older
* Fluent in English

Exclusion Criteria:

For the cluster randomized trial, excluded will be patients who:

* Do not speak English
* Are not Hispanic or Latino(a)
* Have a history of lung cancer
* Had a CT scan in the past 12 months
* Has been coughing up blood in the last two weeks
* Have health conditions that make them poor candidates for curative treatment as determined by the primary care provider,
* Are unable to provide informed consent Interviews

Providers/administrators will be excluded if they:

* Are unable to provide informed consent Online surveys
* Are unable to provide informed consent
* Women who are pregnant.

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 week post-intervention
  The investigators expect a recruitment rate of ≥60%.
Participant Acceptability | 1 week post-intervention
  The Ottawa Acceptability Measure will assess the acceptability of the TELESCOPE intervention from the patient's perspective at 1-week post-intervention. There is no total score for this measure. Responses will be reported descriptively in terms of proportions responding positively or negatively for each criteria.
Follow-up completion rate | 1 week post-intervention
  The investigators expect that ≥90% of Hispanic participants will complete the 1-week follow-up assessments
Intervention Fidelity Rate | 1 week post-intervention
  The investigators expect that ≥80% of the key intervention components will be delivered with 80% fidelity by the patient navigators.

SECONDARY OUTCOMES:
Rate of participants that have completed LDCT | 3 months post-intervention
  The investigators will assess the rates of completion of LDCT at 3 months post-intervention for all participants. This will be abstracted from patients' medical records.
To assess shared decision making quality | 1 week post-intervention
  This will be assessed with the Shared Decision-Making Process Survey (SDM Process_4), which is a 4-item performance measure of the process and outcome of shared decision making. Scores range from 0 to 4, with higher scores indicating a better process.
Feasibility of intervention (Clinicians) | 12 months post-intervention
  The feasibility of the intervention (FIM) measure will be completed by clinicians. The total score for this instrument ranges from 4 to 20, with higher scores indicating greater feasibility.
Clinicians Acceptability | 12 months post-intervention
  The acceptability of the intervention (AIM) will be completed by clinicians. The total score ranges from 4 to 20, with higher scores indicating greater acceptability.
Intervention Appropriateness (Clinicians) | Post-intervention
  The Intervention Appropriateness Measure (IAM) will be completed by clinicians. The total score for each instrument ranges from 4 to 20, with higher scores indicating greater acceptability.

OTHER OUTCOMES:
Tobacco treatment referral | 3 months post-intervention
  Medical records will be reviewed at 3 months post-intervention to determine if a tobacco treatment referral has been generated.
Receipt of tobacco treatment | 3 months post-intervention
  Medical records will be reviewed at 3 months post-intervention to determine if the patient has undergone tobacco treatment.
Cancer Fatalism | Baseline and 1-week post-intervention
  The investigators will assess cancer fatalism by asking participants to rate how much they agree or disagree with 3 items: 1) It seems like everything causes cancer, 2) There's not much participants can do to lower their chances of getting cancer, and 3) There are so many recommendations about preventing cancer, it's hard to know which ones to follow. Response categories for each item are on a four-point scale ranging from strongly agree to strongly disagree. There is no total score for this survey. Responses will be reported descriptively for each question. This measure has shown good internal consistency (Cronbach's alpha = 0.60).
Decisional Conflict | Baseline and 1-week post-intervention
  The Decisional Conflict Scale is a widely used measure of the degree to which a patient feels clear about the options and sure about the choice they make. The scale is scored from 0 to 100, with scores under 25 being associated with implementing decisions, while scores above 37.5 suggest delays in decision making.
Medical Mistrust | Baseline and 1-week post-intervention
  The Medical Mistrust Index is a valid and reliable 7-item self-report measure (Cronbach's alpha = 0.76). Participants are asked to rate their agreement with each of the statements on a 4-point Likert scale, ranging from strongly disagree to strongly agree. Scores range from 7 to 28 with higher scores indicating more mistrust.
Telehealth Patient Satisfaction | 1-week post-intervention
  The investigators will assess patient satisfaction with how the telehealth visit/telephone call with the navigator went for them. Participants are asked 6 questions to determine their perception of the overall quality of their telehealth visit. Response categories for each item are on a 5-point scale ranging from strongly agree to strongly disagree. There is no total score for this survey. Responses will be reported descriptively for each question.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Arana, DrPH, Principal Investigator — Rutgers Cancer Institute of NJ
Locations (1):
- Rutgers Cancer Institute, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No